CLINICAL TRIAL: NCT01535222
Title: A Double-blind, Placebo-controlled, Randomized, Single Ascending Dose Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MDCO-2010 in Patients Undergoing Elective CABG Surgery
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of MDCO-2010 in Patients Undergoing Elective Coronary Artery Bypass Graft Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TMC-CU-10-01
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Results first posted 2012-07-19 (Estimated); Last update posted 2012-07-19 (Estimated); Status verified 2012-06

CONDITIONS: Coronary Artery Bypass Graft; Cardiopulmonary Bypass
Keywords: cardiac surgery; coronary artery bypass graft; cardiopulmonary bypass; haemostasis modulator; blood loss; direct inhibitor of plasmin and plasma kallikrein; CABG; CPB
MeSH Terms: conditions — Hemorrhage | interventions — CU-2010

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Cohort 1 (Experimental): 3 patients: loading dose 0.005 mg/kg; infusion 0.0125 mg/kg/h; pump prime 0.02 mg
  Interventions: Drug: MDCO-2010
- Cohort 2 (Experimental): 3 pts: loading dose 0.011 mg/kg; infusion 0.0250 mg/kg/h; pump prime 0.04 mg
  Interventions: Drug: MDCO-2010
- Cohort 3 (Experimental): 6 patients: loading dose 0.027 mg/kg; infusion 0.0625 mg/kg/h; pump prime 0.09 mg
  Interventions: Drug: MDCO-2010
- Cohort 4 (Experimental): 6 patients: loading dose 0.054 mg/kg; infusion 0.1250 mg/kg/h; pump prime 0.18mg
  Interventions: Drug: MDCO-2010
- Cohort 5 (Experimental): 6 patients: loading dose 0.108 mg/kg; infusion 0.2500 mg/kg/h; pump prime 0.35 mg
  Interventions: Drug: MDCO-2010
- Placebo (Placebo Comparator): 8 patients: commercially available NaCl as matching placebo to MDCO-2010 administered as IV infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MDCO-2010 — MDCO-2010 solution for infusion. Dosage: Pump priming dose; Loading dose infusion over 6 minutes; Maintenance infusion for duration of surgery
  Other Names: CU-2010
  Arms: Cohort 1; Cohort 2; Cohort 3; Cohort 4; Cohort 5
Drug: Placebo — Commercially available NaCl
  Arms: Placebo

SUMMARY:
The purpose of this study is to demonstrate that periprocedural infusion of escalating doses of MDCO-2010 is safe and tolerated in patients undergoing elective CABG surgery, to characterize the single dose pharmacokinetics of MDCO-2010, to investigate the effect of MDCO-2010 on pharmacodynamics (biomarkers of fibrinolysis and coagulation parameters), and to investigate the effect on exploratory clinical endpoints of bleeding, transfusion requirements and reexploration.

DETAILED DESCRIPTION:
This protocol describes a study of the investigational drug MDCO-2010 as a haemostasis modulator in patients undergoing elective Coronary Artery Bypass Graft (CABG) surgery involving a cardiopulmonary bypass (CPB).

Perioperative bleeding is a serious complication that adversely affects the morbidity and mortality of cardiac surgery. To alleviate this complication, prophylactic antifibrinolytic therapies are now widely accepted as a strategy to inhibit excessive fibrinolysis.

MDCO-2010, a synthetic small molecule, is a direct inhibitor of plasmin and plasma kallikrein. Both of these have been implicated with impaired haemostasis. In addition, potent inhibition of coagulation factors Xa, XIa and activated Protein C has been demonstrated. Thus, MDCO-2010 has the potential to mitigate excessive fibrinolysis and thrombin generation during cardiac surgery involving a cardiopulmonary bypass. In particular the latter is supposed to provide additional benefits beyond reducing transfusion requirements.

ELIGIBILITY:
Inclusion Criteria

* Men, aged 18 to 80 years or
* Post-menopausal women, aged up to 80 years. Postmenopausal status defined as ≥ 1 year since last menstruation in women with no medical history of hysterectomy or women with a medical history of bilateral oophorectomy
* Planned elective, isolated primary CABG surgery with more than 1 graft, including the use of cardiopulmonary bypass
* Written informed consent prior to any study-related procedure not part of normal medical care

Exclusion Criteria

Patients may not meet any of the following exclusion criteria:

* Planned concomitant surgery including atrial septal defect (ASD) repair, valve replacement, carotid endarterectomy, aortic surgery, any combined procedure or any repeat sternotomy
* Planned Off-pump CABG
* Body weight < 55 kg or > 110 kg
* Planned hypothermia < 28°C
* Major surgical procedures within 30 days of entry
* Placement of drug-eluting stent (DES) within 12 months or of bare-metal stent (BMS) within 6 weeks of entry in a vessel which is not intended to be grafted
* Ejection fraction < 35%
* Preoperative coagulation abnormalities

  * Platelet count < 100,000/cubic mm, or
  * INR > 1.5 or Quick < 40%, or
  * activated partial thromboplastin time (aPTT) > 1.5 x upper limit of normal (ULN)
* Preoperative Hb < 11 g/dL for male patients or < 10 g/dL for female patients
* Patient refusal to receive donor blood products if necessary
* Administration of thienopyridines within 5 days prior to surgery Administration of warfarin within 5 days prior to surgery
* Administration of tirofiban or eptifibatide within 24 hours or administration of abciximab within 5 days prior to surgery
* Administration of fondaparinux within 24 hours prior to surgery
* Creatinine clearance (calculated using Cockroft-Gault equation) < 60 mL/min
* Planned intraoperative use of tranexamic acid or of ε-aminocaproic acid
* History of stroke or transient ischemic attack within 3 months prior to entry
* Known heparin-induced thrombocytopenia
* Known history of thrombophilia, eg, deep vein thrombosis (DVT) with pulmonary embolism
* Active liver disease
* Any condition requiring chronic immunosuppressive medication
* Receipt of an investigational drug or device 30 days prior to entry
* Any other condition which, in the opinion of the investigator, would prevent a patient's participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lars Englberger, PD Dr. Med., Principal Investigator — Insel Gruppe AG, University Hospital Bern

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1: loading dose 0.005 mg/kg; infusion 0.0125 mg/kg/h; pump prime 0.02 mg
- Cohort 2: loading dose 0.011 mg/kg; infusion 0.0250 mg/kg/h; pump prime 0.04 mg
- Cohort 3: loading dose 0.027 mg/kg; infusion 0.0625 mg/kg/h; pump prime 0.09 mg
- Cohort 4: loading dose 0.054 mg/kg; infusion 0.1250 mg/kg/h; pump prime 0.18mg
- Cohort 5: loading dose 0.108 mg/kg; infusion 0.2500 mg/kg/h; pump prime 0.35 mg
- Placebo: commercially available NaCl as matching placebo to MDCO-2010 administered as IV infusion
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo
Started | 3 | 3 | 7 (Patient randomized but did not meet inclusion/exclusion criteria and did not receive study drug) | 6 | 6 | 8
Completed | 3 | 3 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Inclusion/exclusion | 0 | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 7 | 6 | 6 | 8 | 33
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 1 | 4 | 3 | 3 | 3 | 16
  >=65 years | 1 | 2 | 3 | 3 | 3 | 5 | 17
Age Continuous [Mean (Standard Deviation); unit: years] | 63.3 (12.1) | 62 (10.8) | 59 (8.3) | 68 (9.6) | 63.2 (12.4) | 65.9 (5.6) | 63.9 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 2 | 3 | 0 | 5
  Male | 3 | 3 | 7 | 4 | 3 | 8 | 28
Region of Enrollment [Number; unit: participants]
  Switzerland | 3 | 3 | 7 | 6 | 6 | 8 | 33

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Adverse Events
Description: Number of patients experiencing Adverse Events
Time Frame: 7 days (day of surgery to day 7)
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 8
participants | 3 | 3 | 5 | 4 | 6 | 7

2. Primary Outcome: Incidence of Serious Adverse Events
Description: Number of patients experiencing Serious Adverse Events
Time Frame: 7 days (day of surgery to day 7)
Measure: Number; unit: participants
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo
Number analyzed (Participants) | 3 | 3 | 6 | 6 | 6 | 8
participants | 0 | 0 | 1 | 0 | 2 | 0

ADVERSE EVENTS:
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 1/6 | 0/6 | 2/6 | 0/8
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 5/6 | 4/6 | 6/6 | 7/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=6) | Cohort 4 (N=6) | Cohort 5 (N=6) | Placebo (N=8)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device leakage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=3) | Cohort 3 (N=6) | Cohort 4 (N=6) | Cohort 5 (N=6) | Placebo (N=8)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Chest pain (General disorders) | 2 (2) | 2 (2) | 3 (3) | 1 (1) | 1 (1) | 4 (4)
Post procedural MI (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Alanine aminotransferase (ALAT) increased (Investigations) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 2 (2)
Aspartate aminotransferase (ASAT) increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3) | 3 (3)
Blood creatine phosphokinase MB increased (Investigations) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor can review results communications prior to public release. Sponsor will complete review within 60 days. If Sponsor believes proposed publication contains patentable information, disclosure shall be delayed to 90 days to permit patent filing. If additional time is required an extension shall be granted not to exceed an additional 90 days. If Sponsor believes proposed publication contains confidential information, site shall delete such information.